CLINICAL TRIAL: NCT06992271
Title: A Novel Eccentric Resistance Training Strategy to Maximize Exercise Induced Muscle Damage in Young Adults
Brief Title: Comparing Two Eccentric Protocols on Muscle Damage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BHS-1835
Record Dates: First submitted 2023-03-09; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-11

CONDITIONS: Eccentric Hypertrophy; Muscle Damage

STUDY DESIGN:
Intervention Model Description: Crossover design with two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fast Eccentric (Experimental): Participants will perform fast eccentric resistance training
  Interventions: Behavioral: Fast Eccentric
- Slow eccentric (Active Comparator): Participants will perform slow eccentric resistance training
  Interventions: Behavioral: Slow Eccentric

INTERVENTIONS:
Behavioral: Fast Eccentric — Resistance training done quickly
  Arms: Fast Eccentric
Behavioral: Slow Eccentric — Resistance training done slowly
  Arms: Slow eccentric

SUMMARY:
The purpose of this study will be to test whether a new way of weight training is more effective than typical weight training. The investigators expect that this new way will cause more exercise-induced muscle damage, which helps people build bigger muscles. Another purpose of this study will be to explore perceptions of how muscle soreness impacts participant activities of daily living.

DETAILED DESCRIPTION:
Participants will come to the lab for 3 sessions, plus two email follow-up questionnaires.

Session 1 (45 minutes)

* Complete a demographic questionnaire
* Self-assess muscle soreness
* Walk on the treadmill to warm-up
* Maximal voluntary contraction on the chest press
* Two sets of eccentric (lowering) bench press at 75% of max

Session 2 (45 minutes)

* Walk on the treadmill to warm up
* Maximal voluntary contraction on the chest press
* Three sets of 10 eccentric contractions at 75% of max
* Repeat the maximal voluntary contraction on the chest press

Session 2 Follow-up Rate muscle soreness for each of the three days following Session 2 Answer open-ended questions about perceptions of the muscle soreness

Session 3 (45 minutes) Walk on the treadmill to warm up Maximal voluntary contraction on the chest press Three sets of 10 eccentric contractions at 75% of max Repeat the maximal voluntary contraction on the chest press

Session 3 Follow-up Rate muscle soreness for each of the three days following Session 2 Answer open-ended questions about perceptions of the muscle soreness

ELIGIBILITY:
Inclusion Criteria:

* Sixteen young adults (ages 18-35) will be enrolled in this study.
* In order to be enrolled, they must have completed at least three months of resistance training in the past five years in order to minimize the learning effect and chance of injury.

Exclusion Criteria:

* Since regular resistance training reduces the primary outcomes, muscle damage and soreness, individuals who currently participate in chest press resistance training at least once per week will be excluded.
* Individuals who have musculoskeletal injuries in the shoulder, elbow or wrist that preclude pain-free resistance training, or who have underlying uncontrolled cardiovascular complications will also be excluded.
* Women who are pregnant, or may consider becoming pregnant over the subsequent 2 months, will be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Muscle soreness 1 | 1 day
  Visual analog scale as indirect indicator of muscle damage. Scale of 1-5. Higher score = more soreness
Muscle soreness 2 | 2 days
  Visual analog scale as indirect indicator of muscle damage. Scale of 1-5. Higher score = more soreness
Muscle soreness 3 | 3 days
  Visual analog scale as indirect indicator of muscle damage. Scale of 1-5. Higher score = more soreness
Maximal Voluntary Isometric Contraction Change | pre-intervention, immediately after the intervention
  Change in MVIC will be used to indicated muscle damage.

CONTACTS AND LOCATIONS:
Overall Officials: Amerigo Rossi, Ed.D, Principal Investigator — New York Institute of Technology
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No